CLINICAL TRIAL: NCT05910827
Title: A Phase 1b Study to Evaluate HMBD-001 in Combination With Docetaxel With or Without Cetuximab in Participants With Advanced Squamous Non-Small Cell Lung Cancers, and HMBD-001 in Combination With Cetuximab in Participants With Advanced Squamous Cell Cancers
Brief Title: Study of an Anti-HER3 Antibody, HMBD-001, With Docetaxel +/- Cetuximab in Advanced Squamous Non-small Cell Lung Cancers, and HMBD-001 + Cetuximab in Advanced Squamous Cell Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hummingbird Bioscience (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMBD-001-103
Record Dates: First submitted 2023-06-01; First posted 2023-06-20 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Advanced or Metastatic Squamous Non-Small Cell Lung Cancer; Advanced Head and Neck Squamous Cell Carcinoma; Advanced Esophageal Squamous Cell Carcinoma; Cervical Squamous Cell Carcinoma; Advanced Cutaneous Squamous Cell Carcinoma
Keywords: NSCLC; Non-small Cell Lung Cancer; sqNSCLC; Lung; Squamous; HER3; ErbB3; Docetaxel; Cetuximab; cervical squamous cell carcinoma; HNSCC; CSCC; ESCC; advanced squamous cell cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Participants receive HMBD-001 with docetaxel. This treatment arm is closed to recruitment.
  Interventions: Drug: HMBD-001; Drug: Docetaxel
- Arm B (Experimental): Participants receive HMBD-001 with docetaxel plus cetuximab
  Interventions: Drug: HMBD-001; Drug: Docetaxel; Drug: Cetuximab
- Arm C (Experimental): Participants receive HMBD-001 with cetuximab
  Interventions: Drug: HMBD-001; Drug: Cetuximab

INTERVENTIONS:
Drug: HMBD-001 — HMBD-001 is a humanized Immunoglobulin G1 (IgG1) anti-Human Epidermal Growth Factor Receptor 3(HER3) monoclonal antibody (mAb). It is administered intravenously (IV) weekly
Drug: Docetaxel — Docetaxel 75 mg/m^2 or 60 mg/m IV once every 3 weeks
  Arms: Arm A; Arm B
Drug: Cetuximab — Cetuximab 400 mg/m^2 IV loading dose, followed by 250 mg/m^2 weekly
  Arms: Arm B; Arm C

SUMMARY:
This is a phase 1b multi-center, open-label study of HMBD-001 in combination with docetaxel with or without cetuximab in participants with locally advanced or metastatic squamous Non-Small Cell Lung Cancers, and HMBD-001 in combination with cetuximab in participants with advanced Squamous Cell Cancers

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and be willing to sign an informed consent form

  * Males and females aged over 18 years (or having reached the age of majority according to local laws if the age of majority is > 18 years of age)
  * Eastern Cooperative Oncology Group (ECOG) status of 0 to 1
  * Arm B only: Locally advanced or metastatic squamous non-small cell lung cancer for which all available standard of care treatment options have been exhausted or refused and for which at least one lesion is measurable
  * Arm C only: Advanced or metastatic sqNSCLC, HNSCC, ESCC, CSCC or cervical SCC with at least one prior line of systemic therapy,
  * Have an estimated life expectancy of at least 3 months
  * Participants must be willing to provide a fresh tumor biopsy sample
  * Have adequate organ function
  * Females must be non-pregnant and non-lactating, willing to use a highly effective method of contraception from screening until study completion or be either surgically sterile or post-menopausal
  * Males must be surgically sterile, abstinent, or if engaged in sexual relations with a woman of child-bearing potential, the participant and his partner must be surgically sterile or using an acceptable, highly effective contraceptive method from screening until study completion

Exclusion Criteria:

* Prior treatment with HMBD-001, docetaxel, cetuximab or any other agent that targets Epidermal Growth Factor Receptor (EGFR) or HER3, including pan-HER inhibitors. Prior treatment with docetaxel is allowed for Arm C

  * Receipt of prior targeted therapy, including but not limited to those targeting EGFR activating mutations, ALK fusions, ROS rearrangements, RET fusions or mutations, BRAF V600E mutation, MET exon 14 skipping mutation, and/or KRAS G12C mutation
  * Persistent clinically significant toxicities (Grade ≥2) from previous anti-cancer therapy except for Grade >2 toxicities that are considered unlikely to put the participant at an increased risk of treatment-related toxicity and/or impact the study results e.g., alopecia
  * Most recent anti-cancer therapy including radiotherapy at least 4 weeks, or nitrosourea or mitomycin 3 at least 6 weeks, or 5 half-lives whichever is shorter prior to starting the assigned study treatment
  * Symptomatic primary Central Nervous System (CNS) cancer or metastases unless the symptoms are stable for at least 28 days prior to the first dose of the study drug and any symptoms have returned to baseline
  * Evidence of abnormal cardiac function
  * History of uncontrolled allergic reactions and/or known expected hypersensitivity to the study drugs used in the treatment arm to which the participant is to be enrolled into
  * Any other known active malignancy except for treated cervical intraepithelial neoplasia, or non-melanoma skin cancer
  * Any uncontrolled illness or significant uncontrolled condition(s) requiring systemic treatment
  * Known Human Immunodeficiency Virus (HIV) infection
  * Active hepatitis B or hepatitis C infection
  * Pregnant or breast feeding
  * COVID 19 infection within 3 months prior to the first dose of the study drug
  * COVID 19 vaccination within 14 days prior to the first dose of the study drug
  * Treatment with strong inhibitors or inducers of CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Nature of Adverse Events (AEs) | From the time the Informed Consent Form (ICF) is signed until 30 days after last dose of study treatment
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered to be related to the study treatment
Objective Response Rate (ORR) by Response Evaluation Criteria In Solid Tumors (RECIST) V1.1 | Up to 24 months
  The ORR is defined as the proportion of subjects with confirmed Complete Response (CR) or confirmed Partial Response (PR), based on RECIST Version 1.1
Number of participants with dose-limiting toxicities (DLTs) | During the first three weeks of study treatment
  DLTs will be assessed in the dose escalation cohorts and are defined as toxicities that meet pre-defined severity criteria and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle (3 weeks) of treatment

CONTACTS AND LOCATIONS:
Locations (20):
- Australia (8):
  - GenesisCare North Shore, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - ICON Cancer Centre South Brisbane, Brisbane, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Cabrini Health, Malvern, Victoria
  - Linear Clinical Research, Perth, Western Australia
- The Institute of Oncology, ARENSIA Exploratory Medicine Phase I Unit, Chisinau, Moldova
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Taipei Medical University - Shuang Ho Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No